CLINICAL TRIAL: NCT04204408
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Subcutaneous Doses of NNC0365-3769 (Mim8) in Healthy Subjects and in Subjects With Haemophilia A With or Without Factor VIII Inhibitors
Brief Title: A Research Study Investigating Mim8 in People With Haemophilia A
Acronym: FRONTIER1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN7769-4513; U1111-1227-4220 (Other: World Health Organization (WHO)); 2019-000465-20 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Haemophilia A With or Without Inhibitors

STUDY DESIGN:
Intervention Model Description: Part 1 placebo-controlled double-blind within cohorts (phase 1) Part 2 open-label (phase 2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single dose (part 1) Mim8 (Experimental): Blinded. Single doses in healthy volunteers. Dose escalation. In each of the 6 cohorts, 6 participants will receive Mim8.
  Interventions: Drug: NNC0365-3769 (Mim8)
- Single dose (part 1) placebo (Placebo Comparator): Blinded. Single doses in healthy volunteers. In each of the 6 cohorts, 2 participants will receive placebo.
  Interventions: Drug: Placebo (Mim8)
- Multiple dose (part 2) (Experimental): Open-label. There will be 4 cohorts receiving once-weekly doses (part 2 cohorts 1, 2, 3 and 5) and one cohort receiving once-monthly doses (part 2 cohort 4). Participants will continue into the part 2 extension on the same treatment regimen.
  Interventions: Drug: NNC0365-3769 (Mim8)

INTERVENTIONS:
Drug: NNC0365-3769 (Mim8) — Mim8 administered subcutaneously (s.c., under the skin). The treatment period will consist of 12 once-weekly doses or 3 once-monthly doses
  Arms: Multiple dose (part 2); Single dose (part 1) Mim8
Drug: Placebo (Mim8) — Mim8 placebo administered subcutaneously (s.c., under the skin)
  Arms: Single dose (part 1) placebo

SUMMARY:
This study is investigating how Mim8 works in people with haemophilia A, who either have inhibitors or do not have inhibitors. Mim8 is a new medication that will be used for prevention of bleeding episodes. Mim8 works by replacing the function of the missing clotting factor VIII (FVIII). Mim8 will be injected with a thin needle in the skin of the stomach, using a pen-injector.

The study will last for up to 44 months. It consists of a main phase (part 1 and part 2) and an extension phase. In part 1, participants will be injected only once with either Mim8 or a "dummy" medicine (placebo) - which one will be decided by chance. In part 2 and the extension phase participants will get an Mim8 injection weekly or monthly.

ELIGIBILITY:
Inclusion Criteria:

Single ascending dose part 1:

* Male, aged 18-45 years (both inclusive) at the time of signing informed consent
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Multiple ascending dose part 2:

* Male, aged 12-64 years (both inclusive) at the time of signing informed consent (Germany and Japan have local requirements)
* Diagnosis of congenital haemophilia A with FVIII activity below 1% based on medical records

Exploratory biomarker cohort:

* Male, aged equal to or above 12 years at the time of signing informed consent (Germany and Japan have local requirements)
* Diagnosis of congenital haemophilia A with FVIII activity below 1% based on medical recordsv

Exclusion Criteria:

Part 1:

* Factor VIII activity equal to or above 150% at screening
* Increased risk of thrombosis, e.g. known history of personal or first degree relative(s) with unprovoked deep vein thrombosis
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease

Part 2:

* Known congenital or acquired coagulation disorders other than haemophilia A
* Increased risk of thrombosis as evaluated by the investigator. E.g. known history of personal or first degree relative(s) with unprovoked deep vein thrombosis with exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease with exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing
* Advanced atherosclerotic disease (e.g. known history of ischemic heart disease, ischemic stroke) as evaluated by the investigator
* Any autoimmune disease that may increase the risk of thrombosis
* Receipt of emicizumab or drugs with similar modes of action within 5 half-lives before trial product administration
* Ongoing or planned immune tolerance induction therapy

Exploratory biomarker cohort:

* Known congenital or acquired coagulation disorders other than haemophilia A
* Increased risk of thrombosis as evaluated by the investigator. E.g. known history of personal or first degree relative(s) with unprovoked deep vein thrombosis with exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease with exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing
* Advanced atherosclerotic disease (e.g. known history of ischemic heart disease, ischemic stroke) as evaluated by the investigator
* Any autoimmune disease that may increase the risk of thrombosis
* Ongoing or planned immune tolerance induction therapy

Min Age: 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of treatment emergent adverse events | From time of dosing (Day 1) to Week 16
  Count
Part 2: Number of treatment emergent adverse events | From time of first dosing (Day 1) to Week 12
  Count
Part 2, extension: Number of treatment emergent adverse events | From Week 12 up to Week 176 (16 weeks after last dose)
  Count

SECONDARY OUTCOMES:
Part 1: Number of injection site reactions | From time of dosing (Day 1) to Week 16
  Count
Part 1: Relative change in D-dimer | From baseline (Day 1) to Week 16
  Percent
Part 1: Relative change in prothrombin fragment 1 and 2 | From baseline (Day 1) to Week 16
  Percent
Part 1: Relative change in fibrinogen | From baseline (Day 1) to Week 16
  Percent
Part 1: Relative change in platelets | From baseline (Day 1) to Week 16
  Percent
Part 1: Cmax, SD: the maximum concentration of Mim8 after a single dose | From baseline (Day 1) to Week 16
  μg/mL
Part 1: AUC0-inf, SD: the area under the Mim8 concentration-time curve from time 0 to infinity after a single dose | From baseline (Day 1) to Week 16
  μg*day/mL
Part 1: t1/2, SD: the terminal half-life of Mim8 after a single dose | From baseline (Day 1) to Week 16
  Days
Part 1: tmax, SD: the time to maximum concentration of Mim8 after a single dose | From baseline (Day 1) to Week 16
  Days
Part 1: Change in activated partial thromboplastin time | From baseline (Day 1) to Week 16
  Seconds
Part 2 (weekly and monthly dosing): Number of injection site reactions | From time of first dosing (Day 1) to Week 12
  Count
Part 2 (weekly and monthly dosing): Occurrence of anti-Mim8 antibodies | From baseline (Day 1) to Week 12
  Count
Part 2 (weekly and monthly dosing): Relative change in D-dimer | From baseline (Day 1) to Week 12
  Percent
Part 2 (weekly and monthly dosing): Relative change in prothrombin fragment 1 and 2 | From baseline (Day 1) to Week 12
  Percent
Part 2 (weekly and monthly dosing): Relative change in fibrinogen | From baseline (Day 1) to Week 12
  Percent
Part 2 (weekly and monthly dosing): Relative change in platelets | From baseline (Day 1) to Week 12
  Percent
Part 2 PK session 2 (weekly dosing): Cmax, MD: the maximum concentration of Mim8 after multiple doses | From Day 57 to Day 64
  μg/mL
Part 2 PK session 2 (weekly dosing): AUCτ, MD: the area under the Mim8 concentration-time curve in the dosing interval after multiple doses | From Day 57 to Day 64
  μg*day/mL
Part 2 PK session 2 (monthly dosing): Cmax, MD: the maximum concentration of Mim8 after multiple doses | From Day 57 to Day 85
  μg/mL
Part 2 PK session 2 (monthly dosing): AUCτ, MD: the area under the Mim8 concentration-time curve in the dosing interval after multiple doses | From Day 57 to Day 85
  μg*day/mL
Part 2 (weekly dosing): Mean of maximum thrombin generation (peak height) | From Day 57 to Day 64
  nM
Part 2 (monthly dosing): Mean of maximum thrombin generation (peak height) | From Day 57 to Day 85
  nM
Part 2, extension: Number of injection site reactions | From Week 12 up to Week 176 (16 weeks after last dose)
  Count
Part 2, extension: Occurrence of anti-Mim8 antibodies | From Week 12 up to Week 176 (16 weeks after last dose)
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (39):
- United States (15):
  - Arizona H&T Phoenix Child Hosp, Phoenix, Arizona
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Rush University Med. Cntr, Chicago, Illinois
  - University of Iowa_Iowa City, Iowa City, Iowa
  - University Of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - St. Jude Clinic Novant Health, Charlotte, North Carolina
  - Cincinnati Child's Hsp Med Ctr, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children Hemostati Ctr, Dayton, Ohio
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
  - Vanderbilt Hemostasis Thrombosis Clinic, Nashville, Tennessee
  - Versiti, CCBD, Milwaukee, Wisconsin
- Universitätsklinik für Innere Medizin V, Innsbruck, Austria
- UMHAT Tsaritsa Yoanna - ISUL EAD, Pediatric clinical hematology and oncology, Sofia, Bulgaria
- Germany (2):
  - Charité - Campus Charité Mitte - Charité Research Organisation GmbH, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum im Friedrichshain, Berlin
- Italy (2):
  - Istituto di Medicina Int. A. Bianchi Bonomi Univ. Milano, Milan, MI
  - Policlinico Umberto I Sezione Ematologia, Roma
- Japan (3):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Nara Medical University Hospital_Pediatrics, Nara
  - Tokyo Medical Univ. Hospital_Laboratory Medicine, Tokyo
- Poland (3):
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan, Greater Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Szpital Uniwersytecki, Oddzial Kliniczny Hematologii, Krakow
- South Africa (2):
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng
  - Pietersburg Hospital, Polokwane, Limpopo
- Spain (3):
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital La Fe - Hemostasia y Trombosis, Valencia
- Switzerland (2):
  - Universitätsklinik für Hämatologie, Bern
  - Universitätsspital Zürich - Klinik für Medizinische Onkologie und Hämatologie, Zurich
- Turkey (Türkiye) (3):
  - Hacettepe Üniversitesi Hastanesi- Endokrinoloji, Ankara
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Edirne
  - Ege Üniversitesi Hastanesi- Hematoloji, Izmir
- United Kingdom (2):
  - Royal Free Haemophilia Comprehensive Care Centre, London
  - Oxford Haemophilia Comprehensive Care Center, Oxford

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Chowdary P, Lentz SR, Gil L, Lopez-Jaime FJ, Windyga J, Ong Clausen WH, Laursen PN, Mahlangu J. FRONTIER1 multiple ascending dose extension: a safety, tolerability, pharmacokinetics, and pharmacodynamics study of Mim8 in people with hemophilia A. Res Pract Thromb Haemost. 2025 Oct 8;9(7):103207. doi: 10.1016/j.rpth.2025.103207. eCollection 2025 Oct. PMID 41246456